CLINICAL TRIAL: NCT07050823
Title: Case-Finding for Chronic Respiratory Diseases in People Living With Other Long-Term Conditions
Brief Title: Mitigating Chronic Respiratory Disease Through the Lens of Multi-Morbidity
Acronym: MARES1
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Universidade Federal de Sao Carlos (Other)
Responsible Party: Sponsor
Other Study IDs: 6981600; NIHR 303125 (Other Grant/Funding Number: UK NIHR (National Institute for Health and Care Research))
Record Dates: First submitted 2025-06-13; First posted 2025-07-03 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Asthma; Preserved Ratio Impaired Spirometry
Keywords: case-finding; chronic obstructive pulmonary disease; asthma; multi-morbidity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to make it easier to find people with undiagnosed long-term lung health problems (such as asthma, and chronic obstructive pulmonary disease, COPD, collectively called 'Chronic Respiratory Diseases', CRDs) living in Brasil.

Because people with undiagnosed CRDs often have other medical problems too, such as heart problems, high blood pressure and diabetes (collectively called 'Long Term Conditions', LTC), the investigators will look for undiagnosed CRD in people with LTC when they are attending appointments at local health centres in the cities of Sao Carlos and Sao Paulo.

To look for undiagnosed CRDs the investigators will use two questionnaire-based methods called 'COLA' and 'SBQ'. These are quick and simple to do. All participants will also have tests of their lung function completed including spirometry and Fractional Exhaled Nitric Oxide so that the investigators can make a definite diagnosis of CRDs. When the study is complete, the investigators will examine how well the COLA and SBQ questionnaires perform in identifying people with a definite diagnosis of CRD.

In total, the investigators aim to recruit 859 people.

DETAILED DESCRIPTION:
This study aims to evaluate the discriminative capacity of the COLA-6 questionnaire in identifying individuals with chronic respiratory diseases (CRDs) who attend primary health care (PHC) services in Brasil, for the treatment of other long-term conditions (LTCs). To achieve this, the investigators will conduct a cross-sectional observational study enrolling 859 individuals with one or more existing LTCs who are receiving care in PHC services. The COLA-6 questionnaire will be administered, and its results will be compared to gold-standard post-bronchodilator spirometry. The performance of the case-finding tool will be assessed using the area under a receiver operating characteristic (ROC) curve.

This study will be conducted in PHC services, including Basic Health units (BHUs) and Family Health Units (FHUs), located in the municipalities of São Carlos and São Paulo, both situated in the state of São Paulo, Brasil. The municipality of São Carlos has a population of 254,857 inhabitants and a gross domestic product (GDP) of R$55,044.88 per capita, with 34 PHC units. In contrast, São Paulo, the state capital, has a population of 11,451,999 inhabitants and a per capita GDP of R$66,872.84, and is served by 471 PHC units.

Individuals will be recruited from PHC services, including BHUs and FHUs, located in the municipalities of São Carlos and São Paulo, Brasil. Eligible individuals with NCDs will be identified through three main strategies: (1) individuals attending BHUs/FHUs with an established LTC profile (e.g., scheduled consultations or monitoring for hypertension, diabetes, etc.); (2) individuals with LTCs identified by community health agents through proactive outreach; and (3) individuals with LTCs who attend PHC services and become aware of the study through passive recruitment methods such as posters, information shared by staff or other patients, and invitations extended during service days. Additionally, posters containing the research team's contact information will be displayed, and invitations will be extended during service days at the BHUs/FHUs. All recruitment procedures will be conducted in accordance with ethical principles, ensuring the protection of participants' rights to privacy and autonomy.

Data collection will be conducted in a single visit by a member of the UFSCar research team. All eligible participants will provide written Informed Consent prior study procedures. The following procedures will be carried out:

Initial assessment;

Application of case-finding tools questionnaires:

COLA-6 questionnaire; Symptom-Based questionnaire (SBQ); Exhaled fraction of nitric oxide (FeNO) measurement; Spirometry (pre- and post-bronchodilator);

Application of disease-specific questionnaires:

Chronic Airways Assessment Test (CAAT) for all individuals with abnormal spirometry; Asthma Control Questionnaire (ACQ-7) for individuals with isolated or overlapping asthma; provision of basic information on access to downstream healthcare services for diagnosis and treatment of participants identified with abnormal spirometry.

Participants will be classified based on spirometry and FeNO results into two groups, primarily according to the recommendations of the Global Initiative for Chronic Obstructive Lung Disease (GOLD) and the Global Initiative for Asthma (GINA):

Abnormal Spirometry: Includes COPD, asthma, asthma-COPD overlap, PRISm, restriction patterns, asthma-PRISm overlap and asthma-restriction overlap.

Normal Spirometry: Participants without lung function abnormalities.

The sample size calculation was based on the performance of the COLA-6 questionnaire for diagnosing COPD in the investigators' previous GECo study where COPD prevalence was 9.4%. With these assumed values, a minimum sample size of n=859 individuals will allow the investigators to estimate the area under (AUC) the receiver operating characteristic (ROC) curve to within 4.5% (based on a 95% confidence interval). According to prevalence studies for CRDs in Brasil, the investigators calculate the ability to identify approximately N=146 individuals with COPD, N=77 with asthma, and N=86 with Preserved Ratio Impaired Spirometry (PRISm) in this study, therefore an estimated sample of N=309 with abnormal spirometry and N=550 with normal spirometry. The investigators will case-find in more people if the expected prevalence is lower to reach these targets.

The investigators will summarise the demographic, and clinical characteristics of participants overall and by those with normal and abnormal spirometry. Based on spirometry results, the investigators will report the prevalence of COPD, asthma, PRISm and restriction, alone and in combination, with 95% confidence intervals. For the primary analysis, the investigators will calculate the AUC of the ROC curves for COLA-6 compared with the gold standard spirometry diagnosis separately for combined CRDs, asthma, COPD and PRISm. Using the previously published threshold for COLA-6 scores of ≥4, the investigators will also calculate sensitivity, specificity, and negative and positive predictive values. In addition, based on the ROC curve the investigators will identify the COLA-6 score threshold that achieves sensitivity of at least 90%. All estimates will be reported with 95% confidence intervals.

Full ethical approval was obtained from the Ethics Committee of the Federal University of São Carlos and UNISA (reference number: MARES-1: 85805425.4.1001.5504) and UCL as described above.

The MARES project is funded by the UK NIHR (project reference 303125) using UK international development funding from the UK Government to support global health research. The views expressed in this publication are those of the the investigators and not necessarily those of the NIHR or the UK government.

ELIGIBILITY:
Inclusion Criteria:

Attending primary health care services in Brasil.

Diagnosed with one or more existing, non-respiratory long-term conditions such as cardiovascular disease, diabetes or hypertension.

Exclusion Criteria:

Clinically unstable in the past month (defined as worsening symptoms requiring emergency care or hospitalization).

Current pregnancy.

Active pulmonary tuberculosis or undergoing treatment for pulmonary tuberculosis.

Current acute respiratory infection.

Cognitive impairment that prevents understanding of the case-finding questionnaire, defined as MMSE score ≤20.

Contraindications to spirometry.

Declines to participate in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People attending primary care clinics in Brasil for treatment or monitoring of an existing non-respiratory long-term condition, for example cardiovascular disease, diabetes and hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 859 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Discriminative accuracy of the 'COLA' case-finding questionnaire for diagnosis of abnormal spirometry | Baseline: all assessments are conducted at one visit and the discriminative accuracy of the 'COLA' case-finding questionnaire for diagnosis of abnormal spirometry will use the COLA and spirometry data from the single visit.
  The investigators will report the sensitivity, specificity, positive and negative predictive value for the ability of the 'COLA' case-finding questionnaire to identify people with abnormal post-bronchodilator spirometry.

SECONDARY OUTCOMES:
Discriminative accuracy of the 'COLA' case-finding questionnaire for diagnosis of specific patterns of abnormal spirometry | Baseline: all assessments are conducted at one visit and the discriminative accuracy of the 'COLA' case-finding questionnaire for diagnosis of asthma, COPD and PRISm will use the COLA and spirometry data from the single visit.
  The investigators will report the sensitivity, specificity, positive and negative predictive value for the ability of the 'COLA' case-finding questionnaire to identify people with asthma, COPD and PRISm separately.
Discriminative accuracy of the 'SBQ' (symptom based questionnaire) case-finding questionnaire for diagnosis of overall, and specific patterns of abnormal spirometry | Baseline: all assessments are conducted at one visit and the discriminative accuracy of the 'SBQ' case-finding questionnaire for diagnosis of abnormal spirometry will use the SBQ and spirometry data from the single visit.
  The investigators will report the sensitivity, specificity, positive and negative predictive value for the ability of the 'SBQ' (symptom based questionnaire) case-finding questionnaire to identify people with abnormal spirometry, and asthma, COPD, and PRISm separately.

CONTACTS AND LOCATIONS:
Overall Officials: John R Hurst, PhD FRCP, Principal Investigator — University College London Hospitals; Renata G Mendes, DFisio/ PPGFt, Principal Investigator — Federal University of Sao Carlos (UFScar), Brasil
Locations (2):
- Brazil (2):
  - Multiple primary care sites, São Carlos, São Paulo
  - Multiple primary care sites, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided
On completion of the final report we will consider IPD sharing where this is aligned with the ethics permissions and data governance regulations.